CLINICAL TRIAL: NCT04258709
Title: Effect of Antenatal Milk Expression on Breastfeeding Outcomes Among Overweight and Obese Women
Brief Title: PRenatal Video-Based Education and PostPARtum Effects
Acronym: PREPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jill R. Demirci, PhD, RN, IBCLC, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: STUDY19030116; R01HD098186 (NIH)
Record Dates: First submitted 2020-02-03; First posted 2020-02-06 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Breastfeeding
Keywords: antenatal milk expression; antenatal colostrum
MeSH Terms: conditions — Breast Feeding | interventions — methylamphotericin B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Statistician completing final analysis of data will be blinded to group assignment. An unbiased, third party will conduct qualitative interviews.
  Participants, obstetric providers in recruitment clinics, and lactation consultant interventionists will be blinded to outcomes of interest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antenatal Milk Expression (AME) Intervention Group (Experimental): Weekly video interactions (weeks 37-40 of pregnancy) with International Board Certified Lactation Consultants (IBCLCs) to teach and reinforce antenatal milk expression. At-home practice of hand expression and collection of any expressed milk.
  Interventions: Behavioral: AME
- Video-based Infant Care Education Control Group (Active Comparator): Weekly video education (weeks 37-40 of pregnancy) on various topics related to infant care (e.g., safe sleep, car seat safety, etc.).
  Interventions: Behavioral: Video-based infant care education

INTERVENTIONS:
Behavioral: AME — Participants receive education on AME and feedback on technique with a remotely-based IBCLC via live streaming video.
  Arms: Antenatal Milk Expression (AME) Intervention Group
Behavioral: Video-based infant care education — Participants view a standard set of web-based streamed videos addressing evidence-based infant care, unrelated to feeding/breastfeeding.
  Arms: Video-based Infant Care Education Control Group

SUMMARY:
The purpose of this randomized controlled trial is to examine the impact of a remotely-delivered antenatal milk expression (AME) intervention versus an attention control condition on breastfeeding outcomes among a sample of 280 nulliparous, non-diabetic women with pre-pregnancy body mass indices ≥ 25. AME involves milk expression and collection in the third pregnancy trimester and is theorized to address multiple barriers to breastfeeding among women with higher BMI, including impaired breastfeeding self-efficacy, insufficient milk supply (critical period endocrine modulation of milk volume), and early formula supplementation in the context of a medically complex birth (availability of banked antenatal milk).

Participants will be enrolled in their third trimester of pregnancy and allocated into one of two study arms: 1) AME instruction delivered by remote, live International Board Certified Lactation Consultants via an innovative app-based telelactation platform; or 2) an attention control condition (video-based infant care education unrelated to infant feeding). Video-based education for both groups will occur in weekly study visits from 37 to 40 weeks gestation, with women in the intervention group continuing AME 1-2 times per day at home.

Measured outcomes of interest will include short and long-term breastfeeding practices (e.g., breastfeeding duration, exclusivity) and participants' experiences with and perceptions of AME.

DETAILED DESCRIPTION:
The purpose of the PREPARE Trial is to examine the impact of an antenatal milk expression (AME) intervention among women with pre-pregnancy BMI 25 or more on breastfeeding outcomes, including breastfeeding self-efficacy, breastfeeding duration and exclusivity, and perception of insufficient milk supply. Specifically, the investigators will:

1. Determine the effect of the AME intervention on short-term breastfeeding outcomes, including breastfeeding self-efficacy and exclusivity, to two weeks postpartum.
2. Explore the sustained effect of the AME intervention on longer-term breastfeeding duration and exclusivity over the first year postpartum.
3. Examine participants' experiences with and perceptions of AME.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who:

  1. have a pre-pregnancy BMI ≥ 25
  2. are ≥ 18 years
  3. are English-speaking
  4. are 34 0/7-36 6/7 gestational weeks
  5. are nulliparous
  6. intend to/have interest in breastfeeding after birth
  7. are having a singleton pregnancy
  8. plan to receive prenatal care and deliver at select hospital/birth facility systems (access to EMR data)

Exclusion Criteria:

1. contraindications to breastfeeding as specified by the American Academy of Pediatrics
2. history of breast reduction surgery or radiation
3. indication for delivery by 37 weeks gestation
4. gestational or pre-existing diabetes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 280 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Demirci, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw (subject level) and/or aggregate data will be shared with other investigators as requested after: 1) publication of main findings; 2) removal of identifiers that would permit linkages to individual research participants; and 3) removal of variables that could lead to deductive disclosure of the identity of individuals. Any individual requests for data sharing will be executed in collaboration with the University of Pittsburgh Institutional Review Board to ensure strict adherence to policies for protections of human subjects. In addition, at the conclusion of the study, de-identified data will be submitted to the National Institute of Child Health and Development (NICHD) Data Repository to ensure public availability.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the conclusion of the study, after publication of main findings.
Access Criteria: Contact study investigator or NICHD for access to data repository.

REFERENCES:
- [Derived] Demirci JR, Glasser M, Bogen DL, Sereika SM, Ren D, Ray K, Bodnar LM, O'Sullivan TA, Himes K. Effect of antenatal milk expression education on lactation outcomes in birthing people with pre-pregnancy body mass index >/=25: protocol for a randomized, controlled trial. Int Breastfeed J. 2023 Mar 16;18(1):16. doi: 10.1186/s13006-023-00552-6. PMID 36927811

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between September 23, 2020 and October 23, 2023. Recruitment occurred via electronic health record scans of prenatal practices involved in the study for patients who met basic eligibility criteria, who then received study advertisements, health system portal messages, and/or approaches by study staff at a prenatal visit. Other recruitment strategies included social media ads, a university research registry, study flyers at clinical sites, and magazine advertisements.
Pre-assignment Details: Of 539 participants assessed for eligibility, 280 met eligibility criteria, agreed to participate, and were randomized to an interventionist group.
Period: Overall Study
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Started | 140 | 140
Completed | 128 | 134
Not Completed | 12 | 6
Not completed — Lost to Follow-up | 10 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Fetal demise | 0 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Measures with numbers analyzed less than the overall baseline numbers include all participants with data collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group | Total
Number analyzed (Participants) | 140 | 140 | 280
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (4.71) | 31.12 (5.2) | 30.57 (4.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 140 | 280
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity assessed at baseline with n=279 participants' data available
  Participants
    number analyzed (Participants) | 139 | 140 | 279
    Hispanic or Latino | 4 | 5 | 9
    Not Hispanic or Latino | 133 | 134 | 267
    Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race assessed at baseline with n=279 participants' data available
  Participants
    number analyzed (Participants) | 139 | 140 | 279
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 6 | 9 | 15
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 10 | 18 | 28
    White | 111 | 106 | 217
    More than one race | 7 | 5 | 12
    Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 140 | 140 | 280
Married [Count of Participants; unit: Participants] — Population: Marital status assessed at baseline with n=279 participants' data available
  Participants
    number analyzed (Participants) | 139 | 140 | 279
    Married | 105 | 106 | 211
    Living with a partner | 21 | 20 | 41
    Single or separated | 13 | 14 | 27
Education level [Count of Participants; unit: Participants] — Population: Education level assessed at baseline with n=279 participants' data available
  Participants
    number analyzed (Participants) | 139 | 140 | 279
    Associates degree | 9 | 5 | 14
    Bachelor's degree | 43 | 52 | 95
    Completed occupational or vocational program | 6 | 0 | 6
    Graduated from high school/GED | 9 | 13 | 22
    Master's or doctoral degree | 55 | 60 | 115
    Some college, no degree | 15 | 9 | 24
    Unknown | 2 | 1 | 3
Employed at enrollment [Count of Participants; unit: Participants] — Population: Employment status at enrollment assessed at baseline with n=279 participants' data available
  Participants
    number analyzed (Participants) | 139 | 140 | 279
    No | 16 | 20 | 36
    Yes, but on leave until after baby's birth | 6 | 4 | 10
    Yes, with reduced hours | 9 | 14 | 23
    Yes, with the same number of hours as before pregnancy | 106 | 101 | 207
    Unknown/unreported | 2 | 1 | 3
Special Supplemental Program for Women, Infants, and Children (WIC) recipient [Count of Participants; unit: Participants] — Population: WIC status assessed at baseline with n=279 participants' data available
  Participants
    number analyzed (Participants) | 139 | 140 | 279
    Yes, current recipient | 16 | 14 | 30
    No, not a current recipient | 121 | 125 | 246
    Unreported/unknown | 2 | 1 | 3
Infant Feeding Intentions Scale Score at enrollment [Mean (Standard Deviation); unit: units on a scale] — Only items 3-5 included from Infant Feeding Intentions (IFI) Scale, as items 1-2 part of study eligibility (score range 0-12, with higher score indicative of stronger intention to exclusively breastfeed up to 6 months postpartum) Population: Scale administered at baseline with n=276 participants' data available
  units on a scale
    number analyzed (Participants) | 137 | 139 | 276
    (all) | 10.59 (2.07) | 10.40 (2.02) | 10.49 (2.04)
Breastfeeding Self-Efficacy Scale (Short Form) Score Baseline [Mean (Standard Deviation); unit: units on a scale] — Score range 14-70, with higher scores indicative of higher breastfeeding self-efficacy Population: Scale administered at baseline with n=276 participants' data available
  units on a scale
    number analyzed (Participants) | 137 | 139 | 276
    (all) | 45.57 (8.04) | 46.16 (8.43) | 45.87 (8.23)
Iowa Infant Feeding Attitude Scale [Mean (Standard Deviation); unit: units on a scale] — Score range 17-85, with higher scores indicative of more positive breastfeeding attitude Population: Scale administered at baseline with n=276 participants' data available
  units on a scale
    number analyzed (Participants) | 137 | 139 | 276
    (all) | 44.42 (4.26) | 44.19 (4.26) | 44.30 (4.25)
Pre-pregnancy BMI [Count of Participants; unit: Participants] — Population: BMI at enrollment assessed at baseline with n=279 participants' data available
  Participants
    BMI 25.0-29.99: number analyzed (Participants) | 139 | 140 | 279
    BMI 25.0-29.99 | 77 | 76 | 153
    BMI ≥ 30.0: number analyzed (Participants) | 139 | 140 | 279
    BMI ≥ 30.0 | 62 | 64 | 126
Pre-pregnancy BMI (Continuous) [Mean (Standard Deviation); unit: lbs/in^2] — Population: BMI at enrollment assessed at baseline with n=279 participants' data available
  lbs/in^2
    number analyzed (Participants) | 139 | 140 | 279
    (all) | 31.1 (5.69) | 30.8 (5.87) | 31.0 (5.77)

OUTCOME MEASURES:

1. Primary Outcome: Breastfeeding Exclusivity
Description: Whether participant is feeding 100% breast milk at 2 weeks postpartum
Time Frame: 2 weeks postpartum
Population: Only includes participants with breastfeeding data available at 2 weeks postpartum (i.e., participants who completed breastfeeding survey item(s) at 2 weeks); note that some participants do not have 2 week breastfeeding data or 2 week survey data, but went on to complete the study by completing subsequent study timepoints
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 131 | 137
Participants | 67 | 84
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .1200, Chi-squared
Statistical Analysis 2: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .0474, Regression, Logistic; Odds Ratio (OR) = .593, 95% CI 2-sided [.352 to .9907] — Adjusted for race, Iowa Infant Feeding Attitudes Score at baseline, infant gestational age, NICU admission, maternal age at enrollment, WIC enrollment at baseline, maternal pre-pregnancy BMI. This is an adjusted odds ratio

2. Primary Outcome: Breastfeeding Self-efficacy
Description: Score on Breastfeeding Self-Efficacy Scale-SF (score range 14-70, with higher score represents better outcome)
Time Frame: 2 weeks postpartum
Population: Please note that this indicates the number of participants who completed the BSES-SF in its entirety at this timepoint. Some participants may not have completed this portion of the survey due to 1) not completing a survey at this timepoint, or 2) reporting breastfeeding discontinuation at this timepoint, rendering this survey not applicable to their current experiences.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 121 | 126
score on a scale | 48.8 (13.8) | 47.7 (11.9)
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .5201, t-test, 1 sided
Statistical Analysis 2: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .9178, Regression, Linear; Slope = .1399, 95% CI 2-sided [-2.5299 to 2.8098]

3. Secondary Outcome: Number of Participants Exclusively Breastfeeding During Postpartum Hospitalization
Description: This variable was derived from the infant's feeding documentation via Electronic Medical Record. Responses for Breastfeeding Exclusivity were categorized as YES if the infant had been fed only their mother's own breast milk. Responses were categorized as NO if they had received anything other than only their mother's own breast milk (e.g., formula + their own milk, formula only).
Time Frame: Postpartum hospitalization (0-4 days postpartum)
Population: Please note that this indicates the number of participants who are represented here reflect only those who had still been active in the study at this point, exclusive of participants that had withdrawn (either by self or study staff).
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 138 | 137
Participants
  Exclusively breastfeeding | 79 | 76
  Not exclusively breastfeeding | 59 | 61
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .8614, t-test, 1 sided
Statistical Analysis 2: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .7836, Regression, Logistic; Odds Ratio (OR) = 1.0763, 95% CI 2-sided [.6364 to 1.8216]

4. Secondary Outcome: Number of Participants Exclusively Breastfeeding at 2 Weeks Postpartum
Description: This variable derived from participant self-report survey emailed at 2 weeks postpartum. Responses for Breastfeeding Exclusivity were categorized as YES if the infant had been fed only their mother's own breast milk. Responses were categorized as NO if they had received anything other than only their mother's own breast milk (e.g., formula + their own milk, formula only).
Time Frame: 2 weeks postpartum
Population: Please note that this indicates the number of participants who are represented here reflect only those who had still been active in the study at this point, exclusive of participants that had withdrawn (either by self or study staff) or did not complete a survey at this timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 121 | 127
Participants
  Exclusively breastfeeding | 45 | 46
  Not exclusively breastfeeding | 76 | 81
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .9788, Chi-squared
Statistical Analysis 2: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .9119, Regression, Logistic; Odds Ratio (OR) = 1.0307, 95% CI 2-sided [.603 to 1.7067]

5. Secondary Outcome: Number of Participants Exclusively Breastfeeding at 6 Weeks Postpartum
Description: This variable derived from participant self-report survey emailed at 6 weeks postpartum. Responses for Breastfeeding Exclusivity were categorized as YES if the infant had been fed only their mother's own breast milk. Responses were categorized as NO if they had received anything other than only their mother's own breast milk (e.g., formula + their own milk, formula only).
Time Frame: 6 weeks postpartum
Population: Please note that this indicates the number of participants who are represented here reflect only those who had still been active in the study at this point, exclusive of participants that had withdrawn (either by self or study staff) or did not complete a survey at this timepoint (either due to breastfeeding cessation at a prior timepoint or failure to complete the survey).
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 123 | 122
Participants
  Exclusively breastfeeding | 64 | 73
  Not exclusively breastfeeding | 59 | 49
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .2173, Regression, Logistic; Odds Ratio (OR) = .7157, 95% CI 2-sided [.4192 to 1.216]

6. Secondary Outcome: Number of Participants Exclusively Breastfeeding at 12 Weeks Postpartum
Description: This variable derived from participant self-report survey emailed at 12 weeks postpartum. Responses for Breastfeeding Exclusivity were categorized as YES if the infant had been fed only their mother's own breast milk. Responses were categorized as NO if they had received anything other than only their mother's own breast milk (e.g., formula + their own milk, formula only).
Time Frame: 12 weeks postpartum
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 104 | 111
Participants
  Exclusively breastfeeding | 67 | 69
  Not exclusively breastfeeding | 37 | 42
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .5209, Regression, Logistic; Odds Ratio (OR) = .7157, 95% CI 2-sided [.4192 to 1.216]

7. Secondary Outcome: Number of Participants Exclusively Breastfeeding at 6 Months Postpartum
Description: This variable derived from participant self-report survey emailed at 6 months postpartum. Responses for Breastfeeding Exclusivity were categorized as YES if the infant had been fed only their mother's own breast milk. Responses were categorized as NO if they had received anything other than only their mother's own breast milk (e.g., formula + their own milk, formula only).
Time Frame: 6 months postpartum
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 94 | 101
Participants
  Exclusively breastfeeding | 0 | 2
  Not exclusively breastfeeding | 94 | 99

8. Secondary Outcome: Breastfeeding Exclusivity (Categorical)
Description: Categorical outcome indicating proportional range of breast milk feeds during postpartum/birth hospitalization (0-4 days postpartum)
Time Frame: 0-4 days postpartum
Population: Data not collected from the EHR for the study due to reliability concerns
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Breastfeeding Exclusivity (Categorical)
Description: Categorical outcome indicating proportional range of breast milk feeds since infant was born
Time Frame: 2 weeks
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 121 | 127
Participants
  0% breast milk | 0 | 0
  1-74% breast milk | 31 | 25
  75-99% breast milk | 45 | 56
  100% breast milk | 45 | 46
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .4258, Chi-squared
Statistical Analysis 2: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .6246, Regression, Logistic; Odds Ratio (OR) = .8882, 95% CI 2-sided [.5523 to 1.4283]

10. Secondary Outcome: Breastfeeding Exclusivity (Categorical)
Description: Categorical outcome indicating proportional range of breast milk feeds in past week
Time Frame: 6 weeks postpartum
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 123 | 122
Participants
  0% breast milk | 15 | 15
  1-75% breast milk | 28 | 20
  75-99% breast milk | 16 | 14
  100% breast milk | 64 | 73
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .5613, Chi-squared
Statistical Analysis 2: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .2173, Regression, Logistic; Odds Ratio (OR) = .7157, 95% CI 2-sided [.4206 to 1.2178]

11. Secondary Outcome: Breastfeeding Exclusivity (Categorical)
Description: Categorical outcome indicating proportional range of breast milk feeds in past week
Time Frame: 12 weeks postpartum
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 104 | 111
Participants
  0% breast milk | 8 | 8
  1-74% breast milk | 18 | 16
  75-99% breast milk | 10 | 17
  100% breast milk | 68 | 70
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .6291, Chi-squared
Statistical Analysis 2: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .5426, Regression, Logistic; Odds Ratio (OR) = 1.1955, 95% CI 2-sided [.8745 to 1.3931]

12. Secondary Outcome: Breastfeeding Exclusivity (Categorical)
Description: Categorical outcome indicating proportional range of breast milk feeds in past week
Time Frame: 6 months postpartum
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 94 | 101
Participants
  0% breast milk | 13 | 11
  1-74% breast milk | 23 | 28
  75-99% breast milk | 38 | 40
  100% breast milk. | 20 | 22
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .9071, Chi-squared
Statistical Analysis 2: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .9328, Regression, Logistic; Odds Ratio (OR) = 1.0233, 95% CI 2-sided [.7751 to 1.2084]

13. Secondary Outcome: Breastfeeding Self-efficacy
Description: Scores on Breastfeeding Self-Efficacy Scale-SF(score range 14-70, with higher score represents better outcome)
Time Frame: 6 weeks postpartrum
Population: Please note that this indicates the number of participants who completed the BSES-SF in its entirety at this timepoint. Some participants may not have completed this portion of the survey due to 1) not completing a survey at this timepoint, or 2) reporting breastfeeding discontinuation at this timepoint, rendering this survey not applicable to their current experience.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 123 | 122
score on a scale | 49.7 (14.3) | 48.8 (13.1)
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .5548, Regression, Linear; Slope = .8213, 95% CI 2-sided [-1.9161 to 3.5588]

14. Secondary Outcome: Breastfeeding Self-efficacy
Description: Scores on Breastfeeding Self-Efficacy Scale-SF(score range 14-70, with higher score represents better outcome)
Time Frame: 12 weeks postpartum
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 104 | 111
score on a scale | 52.6 (13.9) | 49.7 (14.3)
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .3861, Regression, Linear; Slope = 1.2412, 95% CI 2-sided [-1.5771 to 4.0594]

15. Secondary Outcome: Number of Participants Breastfeeding at Postpartum Hospitalization (0-4 Days Postpartum)
Description: This variable was derived from the infant's feeding documentation via Electronic Medical Record. Responses were categorized as YES for Breastfeeding Duration if they answered that they were still feeding their own breast milk to their infant at each respective timepoint. Please note that responses were still classified as a YES if they were combination feeding (e.g., using their own breast milk along with formula, solids, etc.). Responses were categorized as NO if they had ceased to provide any of their own breast milk to their infant.
Time Frame: Postpartum hospitalization (0-4 days postpartum)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 138 | 138
Participants
  Yes | 138 | 136
  No | 0 | 2
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .4779, t-test, 1 sided

16. Secondary Outcome: Number of Participants Breastfeeding at 2 Weeks Postpartum
Description: Participants were asked what their infant was currently being fed. Responses were categorized as YES for Breastfeeding Duration if they answered that they were still feeding their own breast milk to their infant at each respective timepoint. Please note that responses were still classified as a YES if they were combination feeding (e.g., using their own breast milk along with formula, solids, etc.). Responses were categorized as NO if they had ceased to provide any of their own breast milk to their infant.
Time Frame: 2 weeks postpartum
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 131 | 137
Participants
  Yes | 121 | 127
  No | 10 | 10
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = 1, Chi-squared
Statistical Analysis 2: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .9163, Regression, Logistic; Odds Ratio (OR) = .9508, 95% CI 2-sided [.3669 to 2.4621]

17. Secondary Outcome: Number of Participants Breastfeeding at 6 Weeks Postpartum
Description: as for outcome 16
Time Frame: 6 weeks postpartum
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 123 | 122
Participants
  Yes | 108 | 107
  No | 15 | 15
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .8031, Regression, Logistic; Odds Ratio (OR) = 1.1084, 95% CI 2-sided [.4937 to 2.4882]

18. Secondary Outcome: Number of Participants Breastfeeding at 12 Weeks Postpartum
Description: as for outcome 16
Time Frame: 12 weeks postpartum
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 104 | 111
Participants
  Yes | 96 | 103
  No | 8 | 8
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .8175, Regression, Logistic; Odds Ratio (OR) = 1.1346, 95% CI 2-sided [.3882 to 3.3161]

19. Secondary Outcome: Number of Participants Breastfeeding at 6 Months Postpartum
Description: as for outcome 16
Time Frame: 6 months postpartum
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 94 | 101
Participants
  Yes | 81 | 90
  No | 13 | 11
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .434, Regression, Logistic; Odds Ratio (OR) = .6964, 95% CI 2-sided [.2813 to 1.7241]

20. Secondary Outcome: Number of Participants Breastfeeding at 12 Months Postpartum
Description: as for outcome 16
Time Frame: 12 months postpartum
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 83 | 91
Participants
  Yes | 50 | 51
  No | 33 | 40
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .4968, Regression, Logistic; Odds Ratio (OR) = 1.2533, 95% CI 2-sided [.6534 to 2.4041]

21. Secondary Outcome: Onset of Lactogenesis II
Description: Recall of lactogenesis II in post-birth days
Time Frame: 2 weeks postpartum
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 128 | 133
Participants
  1 day or less | 5 | 5
  2 days | 16 | 15
  3 days | 40 | 38
  4 days | 32 | 40
  More than 4 days | 33 | 31
  Never | 2 | 4
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .9005, Regression, Logistic; Odds Ratio (OR) = 1.0288, 95% CI 2-sided [.659 to 1.6062]

22. Secondary Outcome: Perceived Milk Supply (Continuous)
Description: Score on PIBBS subscale of H & H Lactation Scale measuring perceived infant satisfaction with breast milk received (score range: 5-35, higher score is better outcome)
Time Frame: 2 weeks postpartum
Population: Please note that this indicates the number of participants who completed the H&H Lactation Scale in its entirety at this timepoint. Some participants may not have completed this portion of the survey due to 1) not completing a survey at this timepoint, or 2) reporting breastfeeding discontinuation at this timepoint, rendering this survey not applicable to their current experience.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 121 | 127
score on a scale | 26.5 (7.92) | 27.7 (6.69)
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .127, Regression, Linear; Slope = -1.4018, 95% CI 2-sided [-3.2052 to .4015]

23. Secondary Outcome: Perceived Milk Supply (Continuous)
Description: as for outcome 22
Time Frame: 6 weeks postpartum
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 108 | 107
score on a scale | 26.7 (8.11) | 28.6 (6.89)
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .07, Regression, Linear; Slope = -1.8958, 95% CI 2-sided [-3.9475 to .1559]

24. Secondary Outcome: Perceived Milk Supply (Continuous)
Description: as for outcome 22
Time Frame: 12 weeks postpartum
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 96 | 103
score on a scale | 26.7 (8.11) | 29.6 (6.67)
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .6299, Regression, Linear; Slope = -0.506, 95% CI 2-sided [-2.574 to 1.562]

25. Secondary Outcome: Perceived Milk Supply (Dichotomous)
Description: Endorsement of insufficient milk supply via investigator created item (dichotomous outcome)
Time Frame: 2 weeks postpartum
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 121 | 127
Participants
  Perceived as insufficient | 32 | 28
  Perceived as sufficient | 89 | 99
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .3835, Regression, Logistic; Odds Ratio (OR) = .7573, 95% CI 2-sided [.4029 to 1.4138]

26. Secondary Outcome: Perceived Milk Supply (Dichotomous)
Description: Endorsement of insufficient milk supply via investigator created item (dichotomous outcome)
Time Frame: 6 weeks postpartum
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 108 | 107
Participants
  Perceived as insufficient | 31 | 26
  Perceived as sufficient | 77 | 81
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .459, Regression, Logistic; Odds Ratio (OR) = .784, 95% CI 2-sided [.409 to 1.4912]

27. Secondary Outcome: Perceived Milk Supply (Dichotomous)
Description: Endorsement of insufficient milk supply via investigator created item (dichotomous outcome)
Time Frame: 12 weeks postpartum
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 96 | 103
Participants
  Perceived as insufficient | 22 | 22
  Perceived as sufficient | 74 | 81
Statistical Analysis 1: Comparison: Antenatal Milk Expression (AME) Intervention Group vs Video-based Infant Care Education Control Group; Test type: Superiority; p = .8499, Regression, Logistic; Odds Ratio (OR) = .9338, 95% CI 2-sided [.458 to 1.9039]

28. Secondary Outcome: Number of Participants Commenting on the Impact/Integration of AME During Pregnancy and Utilization of Antenatally Collected Milk During the Postpartum Period
Description: A subset of participants took place in a qualitative assessment via semi-structured interview. Numbers below represent the number of participants who endorsed each of the following categories during their interview: 1) discussing the impact of the study on their pregnancy/postpartum experience, 2) integration of AME into their daily life, and 3) utilization of antenatal milk during the postpartum period
Time Frame: 6 weeks postpartum
Population: Please note that this indicates the number of participants who were invited, agreed to participate, and completed a qualitative interview at 6 weeks postpartum.
Measure: Count of Participants; unit: Participants
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
Number analyzed (Participants) | 31 | 16
Participants
  Impact of/motivation for AME | 11 | 15
  Integration of AME into daily life | 26 | 0
  Utilization of milk collected antenatally | 11 | 0

ADVERSE EVENTS:
Time Frame: From study enrollment at 34-36 weeks of gestation until conclusion of the intervention and conclusion of primary aims data collection at 2 weeks postpartum. Please note that no adverse events were measured after the 2 week postpartum timepoint.
Description: The unit of measurement here is the maternal participant, where a fetal adverse event was noted, it will be included under the maternal participant.
Arm/Group | Antenatal Milk Expression (AME) Intervention Group | Video-based Infant Care Education Control Group
All-Cause Mortality (participants affected / at risk) | 0/139 | 0/139
Serious Adverse Events (participants affected / at risk) | 71/139 | 66/139
Other Adverse Events (participants affected / at risk) | 113/139 | 74/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Antenatal Milk Expression (AME) Intervention Group (N=139) | Video-based Infant Care Education Control Group (N=139)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 8 | 13 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
Fetal distress as indication for delivery via caesarean section (Pregnancy, puerperium and perinatal conditions) | 6 | 9 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
Fetal demise (Pregnancy, puerperium and perinatal conditions) | 0 | 1 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
NICU admission during postpartum hospitalization (Pregnancy, puerperium and perinatal conditions) | 13 | 13 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
Hyperbilirubinemia requiring phototherapy (Pregnancy, puerperium and perinatal conditions) | 8 | 5 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
Reduced fetal movement during/after AME in past week (Pregnancy, puerperium and perinatal conditions) | 1 | 0/0 — Please note that 1 AME group participant was withdrawn by study staff after enrollment due to exclusion criteria upon EHR review. This adverse event was only collected in the AME Intervention Group since IC group participants did not receive AME
Rupture of membranes during AME (Pregnancy, puerperium and perinatal conditions) | 1 | 0/0 — Please note that 1 AME group participant was withdrawn by study staff after enrollment due to exclusion criteria upon EHR review. This adverse event was only collected in the AME Intervention Group since IC group participants did not receive AME
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 27 | 14 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 2 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 | 3 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
Iron transfusion required during postpartum hospitalization (Pregnancy, puerperium and perinatal conditions) | 1 | 0 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
Partial placental abruption (Pregnancy, puerperium and perinatal conditions) | 0 | 2 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
Postpartum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 15 | 11 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
Infant participant requiring resuscitation beyond SDS after delivery (Pregnancy, puerperium and perinatal conditions) | 3 | 7 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
Infant with hyperbilirubinemia requiring monitoring only (Pregnancy, puerperium and perinatal conditions) | 14 | 9 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
Infant with hypoglycemia (Pregnancy, puerperium and perinatal conditions) | 8 | 6 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
Infant with clavicle fracture (Pregnancy, puerperium and perinatal conditions) | 1 | 0 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
Infant with NAS and prolonged hospitalization (Pregnancy, puerperium and perinatal conditions) | 1 | 0 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
Infant with hip dysplasia (Pregnancy, puerperium and perinatal conditions) | 0 | 1 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
In-patient hospitalization (unrelated to AME) (Pregnancy, puerperium and perinatal conditions) | 1 | 0 — Participant admitted to hospital due to motor vehicle accident; 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
IUGR (Pregnancy, puerperium and perinatal conditions) | 2 | 0 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
Postpartum pre-E with SF (Pregnancy, puerperium and perinatal conditions) | 1 | 0 — Please note that 2 participants (1 from each the AME and infant care group) were withdrawn from the study by study staff immediately after enrollment due to exclusion criteria being met upon EHR review.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Antenatal Milk Expression (AME) Intervention Group (N=139) | Video-based Infant Care Education Control Group (N=139)
Oversupply at 2 weeks postpartum (Pregnancy, puerperium and perinatal conditions) | 39/138 | 21/138 — Please note that 4 participants (2 from each group) were withdrawn prior to the 2 week survey, either by self (n=1) or by staff (n=3) and thus were not followed to the 2 week timepoint
Delivery prior to 39 weeks (Pregnancy, puerperium and perinatal conditions) | 39/138 | 31/138 — Please note that 4 participants (2 from each group) were withdrawn prior to 39 weeks gestation, either by self (n=1) or by staff (n=3)
Lactogenesis II onset < 2 days or > 4 days postpartum or no onset (Pregnancy, puerperium and perinatal conditions) | 39/138 | 41/138 — Please note that 4 participants (2 from each group) were withdrawn prior to the 2 week survey, either by self (n=1) or by staff (n=3) and thus were not followed to the 2 week timepoint
Participant reported emotional discomfort or anxiety with AME while on AME interventionist call (Pregnancy, puerperium and perinatal conditions) | 8/138 | 0/0 — 2 AME participants were withdrawn prior to 37 week interventionist call, either by self or staff and received no intervention. These adverse events were only collected in the AME Intervention Group since IC group participants did not receive AME
Participant reported hand fatigue/pain/discomfort with AME while on AME interventionist call (Pregnancy, puerperium and perinatal conditions) | 6/138 | 0/0 — 2 AME participants were withdrawn prior to 37 week interventionist call, either by self or staff and received no intervention. These adverse events were only collected in the AME Intervention Group since IC group participants did not receive AME
Participant reported breast/nipple discomfort associated with AME while on AME interventionist call (Pregnancy, puerperium and perinatal conditions) | 7/138 | 0/0 — 2 AME participants were withdrawn prior to 37 week interventionist call, either by self or staff and received no intervention. These adverse events were only collected in the AME Intervention Group since IC group participants did not receive AME
Participant reported breast or nipple pain or soreness via daily text diaries (Pregnancy, puerperium and perinatal conditions) | 32/138 | 0/0 — 2 AME participants were withdrawn prior to 37 week interventionist call, either by self or staff and received no intervention. These adverse events were only collected in the AME Intervention Group since IC group participants did not receive AME
Participant reported hand fatigue/hand cramping via daily text message diaries (Pregnancy, puerperium and perinatal conditions) | 25/138 | 0/0 — 2 AME participants were withdrawn prior to 37 week interventionist call, either by self or staff and received no intervention. These adverse events were only collected in the AME Intervention Group since IC group participants did not receive AME
Participant reported anxiety/uneasiness/embarrassment via daily text message diaries (Pregnancy, puerperium and perinatal conditions) | 16/138 | 0/0 — 2 AME participants were withdrawn prior to 37 week interventionist call, either by self or staff and received no intervention. These adverse events were only collected in the AME Intervention Group since IC group participants did not receive AME
Participant reported cramping via daily text message diary (Pregnancy, puerperium and perinatal conditions) | 2/138 | 0/0 — 2 AME participants were withdrawn prior to 37 week interventionist call, either by self or staff and received no intervention. These adverse events were only collected in the AME Intervention Group since IC group participants did not receive AME
Participant reported pelvic pain during daily text message diaries (Pregnancy, puerperium and perinatal conditions) | 1/138 | 0/0 — 2 AME participants were withdrawn prior to 37 week interventionist call, either by self or staff and received no intervention. These adverse events were only collected in the AME Intervention Group since IC group participants did not receive AME
Participant reported lightheadedness/nausea during expression via daily text message diary (Pregnancy, puerperium and perinatal conditions) | 1/138 | 0/0 — 2 AME participants were withdrawn prior to 37 week interventionist call, either by self or staff and received no intervention. These adverse events were only collected in the AME Intervention Group since IC group participants did not receive AME
Participant reported no/little milk output via daily text message diaries (Pregnancy, puerperium and perinatal conditions) | 4/138 | 0/0 — 2 AME participants were withdrawn prior to 37 week interventionist call, either by self or staff and received no intervention. These adverse events were only collected in the AME Intervention Group since IC group participants did not receive AME

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT04258709/Prot_SAP_001.pdf
  • Informed Consent Form (2024-11-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT04258709/ICF_002.pdf